CLINICAL TRIAL: NCT00527956
Title: Facilitation and Barriers to Breastfeeding in the NICU
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: PSY 07-009
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Breastfeeding; Prematurity
Keywords: Breastfeeding premature infants
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To date, there is a paucity of research focusing on maternal breastfeeding goals, how these goals may change after an unexpected event such as a preterm birth, and how mothers of ill and preterm infants define breastfeeding success. No studies were identified that focused exclusively on the breastfeeding goals of mothers of hospitalized preterm infants

The purpose of this study is to answer the following research questions: 1) What are the breastfeeding goals of mothers with preterm infants in the NICU? and 2) What are mothers' perceptions of facilitators and barriers to meeting their breastfeeding goals in the NICU?

DETAILED DESCRIPTION:
As the objective of this study is to describe the breastfeeding goals of mothers and their perceptions of breastfeeding support in the NICU, this study will follow a descriptive, qualitative design. Mothers of preterm newborns in the Royal Victoria Hospital will participate in a semi-structured interview about their breastfeeding goals and what they perceived to be facilitators and barriers to achieving their intended goals. During the interviews, the mothers will be asked a set of socio-demographic questions, open-ended questions about their breastfeeding goals, and open-ended questions about their perceptions of barriers and facilitators to meeting these goals in the NICU Participants may also receive one follow-up phone call to clarify their responses to the questions or to validate the information obtained from the interview.

ELIGIBILITY:
Inclusion Criteria:

1. have one (or more) infant(s) currently admitted in the NICU at the RVH;
2. intended to provide breast milk to their infant(s);
3. are able to speak English; and
4. are willing to be audiotaped during the interview.

Exclusion Criteria:

Include mothers who:

1. never intended to breastfeed;
2. have high risk social situations (for example, known maternal mental illness; involvement of youth protection; known alcohol and drug abuse; adoption; identified congenital anomalies);
3. gave birth at term; and
4. have infants with significant birth defects or serious medical conditions in addition to prematurity.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2007-09; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Ciofani, RN, M.Sc.(A), Principal Investigator — McGill Univsersity Health Centre